CLINICAL TRIAL: NCT01326676
Title: PESCA - A Randomised Controlled Trial of a Cardiovascular Polypill Treatment Strategy Compared With Usual Care on Carotid Intima-media Thickness in Individuals at High Risk of Cardiovascular Disease
Brief Title: Polypill Effects on Sub Clinical Atherosclerosis (PESCA) Trial
Acronym: PESCA
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding never attained
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Royal College of Surgeons, Ireland (Other); UMC Utrecht (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRO1656 (Sub-study of 241849 )
Record Dates: First submitted 2011-03-29; First posted 2011-03-31 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cardiovascular Disease
Keywords: Polypill; Red Heart Pill; Cardiovascular disease; Secondary prevention; carotid intima media thickness
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- polypill (Experimental): Red Heart Pill Version 1 and Red Heart Pill Version 2.
  Interventions: Drug: Polypill: Red Heart Pill
- usual medication (Active Comparator): participants continuing to receive cardiovascular disease medications as separate tablets prescribed by their usual physician
  Interventions: Drug: Usual medication

INTERVENTIONS:
Drug: Polypill: Red Heart Pill — The polypill will be taken once/day in the form of a hard capsule, to be taken orally. There are two versions of the polypill (Red Heart Pill):
  Version 1 contains aspirin 75mg, simvastatin 40mg, Lisinopril 10mg and Atenolol 50mg; Version 2 contains aspirin 75mg, simvastatin 40mg, Lisinopril 10mg and Hydrochlorothiazide 12.5mg.
  Red Heart Pill Version 1 and Red Heart Pill Version 2. In general, participants with a history of coronary heart disease will be given version 1, and those with a history of stroke or cerebrovascular disease will be given version 2.
  Arms: polypill
Drug: Usual medication — Participants in the 'Usual Care' arm will continue to take the separate, individual medications prescribed by their usual doctor, e.g. aspirin, blood pressure lowering drugs, statins.
  Other Names: Usual cardiovascular disease prevention medication
  Arms: usual medication

SUMMARY:
Medications that lower blood pressure and cholesterol are known to improve the shape and function of our blood vessels. These improvements include a reduction in the thickness of the wall of the carotid artery (the main artery that runs up the neck to supply the brain) and a reduction in the stiffness of arteries generally including the main central artery -the aorta. Such medications are in the polypill (the Red Heart Pill) that is being used in the UMPIRE Study. In UMPIRE, patients' reported adherence to taking the single, once daily polypill is being compared to adherence to medications taken as separate tablets (usual care).The aim of the PESCA sub-study is to see whether or not the polypill differs from 'usual care' in its direct effects on blood vessels as shown by ultrasound examination of the carotid arteries and assessment of central (aortic) blood pressure.

DETAILED DESCRIPTION:
PESCA is a substudy of the UMPIRE clinical trial which is evaluating a 'polypill' treatment strategy for subjects with established cardiovascular disease or at high risk. All PESCA subjects will have already been recruited to UMPIRE and randomised to taking either a single 'polypill' (comprising low dose aspirin, a cholesterol-lowering statin, and one of two blood pressure lowering medicines) or their usual treatment consisting of similar medication in more than one separate tablets.

PESCA will evaluate whether: 1) progression of atherosclerosis (fatty deposits which narrow the arteries and impair blood flow to vital organs); and 2) central systolic blood pressure (the pressure in the body's main artery, the aorta, when the heart pumps out blood), are reduced in 'polypill' recipients compared to those who continue their usual treatment. Atherosclerosis and central blood pressure are both strongly associated with increased risk of heart attacks and stroke. Atherosclerosis will be assessed by ultrasound scanning of the carotid (neck) arteries to look at thickness of the artery walls (carotid intima media thickness)and plaques(fatty deposits). Direct measurement of central blood pressure is impractical but it will be estimated using a computerised "pulsecor" device. This uses an inflatable cuff on the arm but provides a detailed recording of the pressure wave as the cuff is deflated which enables "pulsecor" to calculate central blood pressure. Results from both ultrasound and blood pressure investigations will be reviewed by investigators who do not know whether the subjects have been randomised to the polypill or their usual treatment.

PESCA assessments will be conducted at 2 visits:baseline (as soon as possible after recruitment to the UMPIRE study); and at the end of both studies (which will coincide).

Parallel studies are being undertaken in the three European sites (UK, Eire and Netherlands) participating in the UMPIRE trial with each site aiming to recruit 300 participants.

ELIGIBILITY:
Patients must meet the inclusion criteria for the UMPIRE trial, and be consented to take part in the PESCA sub-study.

Inclusion criteria

Individuals are eligible for inclusion if all of the following criteria are satisfied:

Adults (≥ 18 years) The participant is able to give informed consent. Established atherothrombotic cardiovascular disease (CVD) or high cardiovascular risk, defined as;

* History of coronary heart disease (myocardial infarction, stable or unstable angina pectoris, or coronary revascularisation procedure), or
* History of ischaemic cerebrovascular disease (ischaemic stroke or transient ischaemic attack), or
* History of peripheral vascular disease (peripheral revascularisation procedure or amputation due to vascular disease), or
* For individuals without established cardiovascular disease, a calculated 5 year CVD risk of 15% or greater (calculated using the 1991 Anderson Framingham risk equation with adjustments as defined by the New Zealand Guidelines Group recommendations) The trial Investigator considers that each of the polypill components are indicated at the doses in the Red Heart Pill The trial Investigator is unsure as to whether a polypill-based strategy or usual care is better.

Exclusion criteria

Individuals will NOT be eligible if one or more of the following criteria are satisfied:

* Contraindication to any of the components of the polypill (e.g. known intolerance to aspirin, statins, or ACE inhibitors; pregnancy or likely to become pregnant or breastfeeding women during the treatment period).
* The treating doctor considers that changing a participant's cardiovascular medications would put the participant at risk (e.g. symptomatic heart failure, high dose β-blocker required to manage angina or for rate control in atrial fibrillation, accelerated hypertension, severe renal insufficiency, a history of severe resistant hypertension).

Other potential reasons for exclusion include:

* Known situation where medication regimen might be altered for a significant length of time, e.g. current acute cardiovascular event, planned coronary bypass graft operation.
* Unlikely to complete the trial (e.g. life-threatening condition other than cardiovascular disease) or adhere to the trial procedures or attend study visits (e.g. major psychiatric condition, dementia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02 (Estimated); Primary Completion 2012-07 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
change in intima-media (artery wall) thickness in the common carotid artery | from baseline to end of trial follow up (1-2 years)
change in intima-media (artery wall) thickness and extent of atherosclerotic plaques in the carotid artery bifurcation | from baseline to end of trial follow-up (1-2 years)
change in central aortic blood pressure | from baseline to end of trial follow-up (1-2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Simon McG Thom, Principal Investigator — Imperial College London; Alice Stanton, Principal Investigator — Royal College of Surgeons in Ireland; Michiel Bots, Principal Investigator — UMC Utrecht; Alun Hughes, Principal Investigator — Imperial College London
Locations (3):
- Royal College of Surgeons of Ireland Research Institute, Dublin, Ireland
- University Medical Centre Utrecht, Utrecht, Netherlands
- Imperial College London, London, United Kingdom